CLINICAL TRIAL: NCT02465931
Title: Decisional Capacity and Informed Consent in Fragile X Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FXS; 1R01HD071987-01A1 (NIH)
Record Dates: First submitted 2015-05-22; First posted 2015-06-09 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Fragile X Syndrome (FXS)
Keywords: Informed Consent; Fragile X Syndrome; Tablets; Decisional Capacity
MeSH Terms: conditions — Fragile X Syndrome | interventions — Paper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison Condition (Other): Paper and pencil informed consent
  Interventions: Other: Paper and Pencil Informed Consent
- Intervention condition (Experimental): Digital informed consent tool
  Interventions: Other: Digital Informed Consent Tool

INTERVENTIONS:
Other: Paper and Pencil Informed Consent — Paper-based informed consent form will be sent to participant and family before data collection visit. They will be able to review as many times as they wish before visit. During visits, simplified overview of informed consent form will be provided in person just once. For MacArthur Competence Assessment Tool (MacCAT) Questions, All questions will be asked after the disclosure information has been presented. Questions will have the same wording as experimental condition. Procedures will mimic MacCAT/flipchart (incorrect or partial credit will be given opportunity to answer question again after disclosure information is repeated). There will be multiple choice options rather than open-ended. Finally, data collection will be done through paper and pencil.
  Arms: Comparison Condition
Other: Digital Informed Consent Tool — Paper informed consent form will be sent to participant and family before data collection visit. They will be able to review as many times as they wish before visit. During visits, the participant can go through the tablet-based tool up to 3 times. All questions will be embedded within the vignettes/presentation of disclosure information. Question will use simplified wording, similar to flipchart. Procedures will mimic MacArthur Competence Assessment Tool (MacCAT) /flipchart (incorrect or partial credit will be given opportunity to answer question again after disclosure information is repeated). Multiple choice options will be utilized rather than open-ended. Finally, response data stored within tool and exported to dataset for analysis.
  Arms: Intervention condition

SUMMARY:
The Decisional Capacity and Informed Consent in Fragile X Syndrome (FXS) project is for the Eunice Kennedy Shriver National Institute of Child Health & Human Development, 1R01HD071987-01A1, and will provide the first comprehensive description of decisional capacity of individuals with FXS; identify individual, family, and experiential factors associated with variability in decisional capacity; determine the validity of caregiver and expert ratings; and develop evidence-based guidelines for categorizing decisional capacity of individuals with FXS. The researchers will develop a methodologically rigorous and conceptually grounded decision aid using digital technology to enhance participation of individuals with FXS in the consent process.

DETAILED DESCRIPTION:
FXS is the most common inherited form of intellectual disability (ID). The typical male has an IQ (intelligence quotient) of 50 to 55, but involvement ranges from mild to severe. Females are generally less affected and have a broader range in function. Some have severe ID and adaptive impairments, but most have a normal or borderline intellectual ability. This wide range in cognitive skills leads to variable ability to make choices and live independently. Most research on individuals with FXS has been noninvasive, limited to parent surveys and psychological assessments. Studies such as these evoke few if any major ethical concerns, so the consent process typically involves a straightforward parental consent. Some studies have drawn blood, collected saliva, measured heart rate, or used neuroimaging, but until recently there has been a paucity of treatment research. This scenario has changed dramatically in the past several years. Advances in understanding the molecular basis of FXS have led to a new generation of treatments, and clinical trials are under way using a variety of compounds. The possibility of side effects and the potential for significant changes in behavior and ability elevate to a new level the importance of obtaining meaningful consent, not only from parents, but also from individuals with FXS. Researchers and Institutional Review Board (IRB) members need data to guide decisions about involving individuals with FXS in the consent process. Unfortunately, little is known about the extent to which individuals with FXS can be or are involved in decisions about research participation. This project will assess the range of decisional capacity in FXS, identify factors associated with individual differences in decisional capacity, validate a rating scale for categorizing decisional capacity, and develop a novel tablet-based decision aid technology to assist researchers and clinicians in maximizing decisional capacity and consent. This study will work toward achieving two overarching aims: 1) Characterize and explain individual differences in decisional capacity in FXS, 2) Design and evaluate the effect of a tablet-based decision aid on participation in the consent process for a hypothetical clinical trial. Ultimately, this study will provide important information about the nature of decisional capacity in FXS and validate a novel intervention to maximize successful participation in the consent process.

ELIGIBILITY:
Inclusion Criteria:

* Places in the first 3 categories of the MacCAT flip chart
* Can provide informed consent using a standard practice

Exclusion Criteria:

* Not in the first 3 categories of the MacCAT flipchart
* Not able to provide informed consent without significant modifications to consent procedures

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Furberg, PhD, Study Director — RTI International
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furberg RD, Raspa M, Wheeler AC, McCormack LA, Bailey DB. A Digital Health App to Assess Decisional Capacity to Provide Informed Consent: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Nov 19;7(11):e10360. doi: 10.2196/10360. PMID 30455171
- [Derived] Furberg RD, Ortiz AM, Moultrie RR, Raspa M, Wheeler AC, McCormack LA, Bailey DB Jr. A Digital Decision Support Tool to Enhance Decisional Capacity for Clinical Trial Consent: Design and Development. JMIR Res Protoc. 2018 Jun 6;7(6):e10525. doi: 10.2196/10525. PMID 29875084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through research registries and convenience samples
Pre-assignment Details: 41 participants were excluded because they did not meet eligibility criteria
Period: Overall Study
Arm/Group | Intervention Condition | Comparison Condition
Started | 55 | 56
Completed | 44 | 45
Not Completed | 11 | 11
Not completed — Lost to Follow-up | 9 | 11
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Condition | Comparison Condition | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 18 | 35
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.16 (7.11) | 21.27 (7.50) | 21.21 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 17 | 20 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 43 | 44 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 38 | 40 | 78
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 44 | 45 | 89
Stanford Binet 5 verbal IQ (intelligence quotient) score [Mean (Standard Deviation); unit: scores on a scale] — The verbal IQ score of the Stanford Binet 5 provides a composite of all the cognitive skills required to solve the items in the five verbal subtests: fluid reasoning, knowledge, quantitative reasoning, visual-spatial processing, and working memory. The verbal IQ subtests are summed but because individuals with intellectual and developmental disabilities have floor effects on many standardized tests, a z-transformation was used (see Sansone et al. 2014). Unit of measure is the z-transformed verbal IQ score. The range was 40.49 to 110.64 in this sample. A higher score indicates higher verbal IQ.
  scores on a scale | 65.67 (17.26) | 69.48 (16.37) | 68.2 (17.8)

OUTCOME MEASURES:

1. Primary Outcome: Decisional Capacity - Understanding Score
Description: MacArthur Decisional Capacity - understanding score, range 0 (no understanding) to 26 (perfect understanding) A summary score was calculated, ranging from 0-26. Scores were then translated into a percentage based on the number of questions answered. A score of 100% indicates that the participant answered each understanding question correctly on the first attempt.
Time Frame: Day 1, immediately following presentation of the material in the intervention or comparison condition
Measure: Mean (Standard Deviation); unit: percentage of understanding
Arm/Group | Intervention Condition | Comparison Condition
Number analyzed (Participants) | 44 | 45
percentage of understanding | 74.4 (27.3) | 75.1 (25.9)
Statistical Analysis 1: Comparison: Intervention Condition vs Comparison Condition; Test type: Other; p = 0.89, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Day 1, immediately following the presentation of the material in the intervention or comparison condition.
Arm/Group | Intervention Condition | Comparison Condition
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/45
Other Adverse Events (participants affected / at risk) | 0/44 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02465931/Prot_SAP_000.pdf